CLINICAL TRIAL: NCT06430385
Title: A Phase 1-2, Double-Blind, Sham-Controlled Multiple Ascending Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intrathecally-Administered ION440 in Patients With MECP2 Duplication Syndrome
Brief Title: ATTUNE: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intrathecally-Administered ION440 in Participants With Methyl CpG Binding Protein 2 (MECP2) Duplication Syndrome (MDS)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ION440-CS1; 2023-507192-22 (EudraCT Number); U1111-1303-4105 (Other: WHO Number)
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Methyl CpG Binding Protein 2 (MECP2) Duplication Syndrome
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: ION440 Dose A (Experimental): Participants will receive ION440 intrathecally at Dose A during Part 1/MAD, followed by ION440 Dose A during Part 2/LTE.
  Interventions: Drug: ION440
- Cohort 2: ION440 Dose B (Experimental): Participants will receive ION440 intrathecally at Dose B during Part 1/MAD, followed by ION440 Dose B during Part 2/LTE.
  Interventions: Drug: ION440
- Cohort 3: ION440 Dose C (Experimental): Participants will receive ION440 intrathecally at Dose C during Part 1/MAD, followed by ION440 Dose C during Part 2/LTE.
  Interventions: Drug: ION440
- Sham Procedure (Sham Comparator): During the Part 1/MAD period, a lumbar procedure (LP) will be performed at the same frequency as ION440 administration. Participants will not receive ITB injections during this period. It will be followed by the open-label Part 2/LTE period, where participants will receive ION440 at the same dose as their enrolled cohort (e.g. Dose A, Dose B or Dose C).
  Interventions: Procedure: Sham procedure

INTERVENTIONS:
Drug: ION440 — ION440 will be administered by intrathecal bolus (ITB) injection.
  Arms: Cohort 1: ION440 Dose A; Cohort 2: ION440 Dose B; Cohort 3: ION440 Dose C
Procedure: Sham procedure — An LP will be performed with CSF collection but will not be followed by the administration of study treatment by ITB injection.
  Arms: Sham Procedure

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of ION440.

DETAILED DESCRIPTION:
This is a phase 1-2 randomized, double-blind, sham-controlled, multiple-ascending dose (MAD) study to evaluate ION440 in pediatric and adult participants with MECP2 Duplication Syndrome (MDS) and will be conducted in two parts. During Part 1 (MAD) (36 weeks), participants will be randomized in a 3:1 ratio to receive ION440 or sham. Individuals who complete Part 1 may enter Part 2, an open label long-term extension study (LTE), where they will receive ION440 for up to approximately 156 weeks. Multiple dose cohorts (Dose A, Dose B, and Dose C) will be evaluated in the study.

All dosing cohorts will be further subdivided by age. Sub cohort A will include participants 8 through 65 years of age, and sub cohort B will include participants 2 through 7 years of age. Dosing cohorts will be enrolled sequentially with sub cohort A initiating prior to sub cohort B.

ELIGIBILITY:
Key Inclusion criteria for Part 1:

1. Males aged ≥ 2 to ≤ 65 years, depending on specific cohort and group, at the time of informed consent.

   1. Group A: ≥ 8 to ≤ 65 years old
   2. Group B: 2 to 7 years old, inclusive
2. Participant has at least one parent or caregiver ≥ 18 years old capable of providing informed consent and able to comply with all study requirements and activities.
3. Participant has a documented diagnosis of MDS with genetic confirmation of MECP2 duplication.
4. Is currently receiving stable doses of concomitant medications for at least 1 month prior to screening.
5. Able to complete all study procedures, measurements and visits to support primary and secondary endpoints, in the opinion of the Investigator.

Key Exclusion criteria for Part 1:

1. Documented diagnosis of severe MECP2 duplications including terminal duplication and/or translocation or MECP2 triplication OR clinical features associated with severe variant structure including (a) onset of seizures prior to age 5 (for those aged 5 and above at signing of ICF), (b) oxygen dependence, (c) microcephaly, IF MECP2 genetic structure information is unavailable.
2. Clinically significant vital sign or ECG abnormality at Screening
3. Known brain or spinal disease that would interfere with the LP procedure, or CSF circulation or presence of other factors would affect the safety of the LP procedure.
4. Has any concomitant disease or condition or circumstance, or any finding at Screening that, in the opinion of the Investigator, makes the participant unsuitable for enrollment or that could interfere with the conduct of the study or that would pose an unacceptable risk to the participant in this study.
5. Treatment with an investigational drug, biological agent, or device within 30 days of Screening, or 5 half-lives of investigational agent, whichever is longer.
6. Previous treatment with an oligonucleotide (including siRNA) within 4 months of Screening if single dose received, or within 12 months of Screening if multiple doses received (this exclusion does not apply to vaccines - both mRNA and viral vector vaccines are allowed including COVID-19). For centrally administered ASOs, a minimum of 12 months washout is required irrespective of the number of doses received.
7. Currently enrolled in a clinical trial of an investigational agent or device or has used any investigational agent or device within 5 half-lives of investigational agent, whichever is longer.
8. Has a history of gene therapy or cell transplantation or any other experimental brain surgery.
9. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Baseline (Day 1).
10. Has experienced Status Epilepticus in the past 6 months.

Key Inclusion criteria for Part 2:

1. Participants in ION440-CS1, Part 1/MAD who received at least one dose of Study Drug /Sham in Part 1/MAD, missed no more than 1 study visit, and attended the Follow Up visit (Visit 6).
2. All inclusion criteria in Part 1/MAD apply (participants will not be required to undergo new Screening bloodwork).

Key Exclusion criteria for Part 2:

1. Has developed any concomitant disease (e.g., gastrointestinal, renal, hepatic, endocrine, respiratory, or cardiovascular system disease) or condition or circumstance, or any finding during Part 1/MAD that, in the opinion of the Investigator, makes the participant unsuitable for continued treatment (e.g., could interfere with the conduct of the study or that would pose an unacceptable risk to the participant in this study).

Ages: 2 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only males are included for this disease condition.
Enrollment: 48 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Up to approximately 36 weeks
Part 1: Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to approximately 36 weeks
Part 1: Number of Participants With Clinically Significant Change From Baseline in Physical and Neurological Examination Findings | Baseline up to approximately 36 weeks
Part 1: Number of Participants With Clinically Significant Change from Baseline in Laboratory Assessments | Baseline up to approximately 36 weeks
Part 1: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) | Baseline up to approximately 36 weeks
Part 2: Number of Participants With TEAEs | Up to approximately 192 weeks
Part 2: Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to approximately 192 weeks
Part 2: Number of Participants With Clinically Significant Change From Baseline in Physical and Neurological Examination Findings | Baseline up to approximately 192 weeks
Part 2: Number of Participants With Clinically Significant Change from Baseline in Laboratory Assessments | Baseline up to approximately 192 weeks
Part 2: Number of Participants With Clinically Significant Change From Baseline in ECG | Baseline up to approximately 192 weeks

SECONDARY OUTCOMES:
Part 1: Maximum Observed Concentration (Cmax) of ION440 in Plasma | Pre-dose and at multiple points post-dose up to Week 36
Part 1: Area Under the Concentration-time Curve (AUC) of ION440 in Plasma | Pre-dose and at multiple points post-dose up to Week 36
Part 1: Plasma Terminal Elimination Half-life (t½) of ION440 | Pre-dose and at multiple points post-dose up to Week 36
Part 1: Trough Concentration (Ctrough) of ION440 in Plasma and CSF | Pre-dose and at multiple points post-dose up to Week 36
Part 1: Plasma Concentration of ION440 | Pre-dose and at multiple points post-dose up to Week 36
Part 2: Trough Concentration (Ctrough) of ION440 in Plasma and CSF | Up to approximately 192 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- United States (8):
  - Rady Children's Hospital, San Diego, California
  - University of Colorado Hopsital - Anschutz Medical Campus, Aurora, Colorado
  - Kennedy Krieger, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
- Kepler University Hospital, Linz, Austria
- CHU Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/